CLINICAL TRIAL: NCT03755258
Title: A Phase Ib Study to Evaluate the Safety, Efficacy and Pharmacokinetics of GCK in Rheumatoid Arthritis Patients
Brief Title: Trial of Ginsenoside Compound K (GCK) Tablet in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HISUN-GCK-Ib-01
Record Dates: First submitted 2018-11-21; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Early Rheumatoid Arthritis
Keywords: Ginsenoside compound K tablet; Rheumatoid Arthritis; Phase Ib study
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Glucokinase

STUDY DESIGN:
Intervention Model Description: Multiple Ascending Dose, Multiple Groups, Multiple Centers
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GCK 100 mg group (Experimental): GCK 100 mg+ Placebo 200 mg GCK tablet 100 mg + Placebo tablet 100 mgX2 tablets, once daily for 12 weeks (oral)
  Interventions: Drug: GCK 100 mg + Placebo 200 mg
- GCK 200 mg group (Experimental): GCK 200 mg + Placebo 100 mg GCK tablet 100 mg X 2 tablets+ Placebo tablet 100 mg once daily for 12 weeks (oral)
  Interventions: Drug: GCK 200 mg + Placebo 100 mg
- GCK 300 mg group (Experimental): GCK tablet 300 mg GCK tablet 100 mgX3 tablets once daily for 12 weeks (oral)
  Interventions: Drug: GCK 300 mg
- Placebo of GCK group (Placebo Comparator): Placebo 300 mg Placebo tablet 100 mgX3 tablets, once daily for 12 weeks (oral)
  Interventions: Drug: Placebo 300mg

INTERVENTIONS:
Drug: GCK 100 mg + Placebo 200 mg — GCK 100 mg + Placebo 200 mg, oral, 12 weeks
  Other Names: GCK
  Arms: GCK 100 mg group
Drug: GCK 200 mg + Placebo 100 mg — GCK 200 mg + Placebo 100 mg, oral, 12 weeks
  Other Names: GCK
  Arms: GCK 200 mg group
Drug: GCK 300 mg — GCK 300 mg, oral, 12 weeks
  Other Names: GCK
  Arms: GCK 300 mg group
Drug: Placebo 300mg — Placebo 300mg, oral, 12 weeks
  Other Names: Placebo of GCK
  Arms: Placebo of GCK group

SUMMARY:
This is a phase Ib study to investigate the safety, pharmacokinetics and preliminary efficacy of ginsenoside compound K (GCK) tablets in patients with rheumatoid arthritis. This study is to be run in China involving 10-12 sites. It will enroll approximately 240 patients to ensure 128 randomized with active rheumatoid arthritis. The treatment period is 12 weeks and total study duration per patient is approximately 14 weeks.

DETAILED DESCRIPTION:
In this double-blind, placebo-controlled, phase Ib study, 128 patients with active RA are planned to be enrolled and randomly assigned 1:1:1:1 to receive placebo, or different doses of GCK tablet (100/200/300 mg). This study will evaluate the safety, pharmacokinetics and preliminary efficacy of GCK tablets in patients with rheumatoid arthritis

ELIGIBILITY:
Inclusion Criteria:

* Patients have active RA as confirmed by the following criteria:

  1. ≥ 4 swollen joints and ≥ 4 tender joints at screening and baseline using the DAS28 joint count.
  2. ESR ≥ 28 mm/hour, or CRP ≥ 1.5 times ULN.
* Patients on non-prohibited medications must receive stable dose for at least 2 weeks prior to study drug administration and maintain an unchanged regimen during the study.
* Patients who are able and wish to sign the informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

* Patients have prior exposure to any csDMARDs or bDMARDs.
* Patients have received corticosteroids, or Chinese medicine preparations such as tripterygium wilfordii, total glucosides of paeony for RA treatment.
* Patients with fibromyalgia
* Patients diagnosed with any systemic inflammatory disease other than RA, including but not limited to juvenile chronic arthritis, spondyloarthropathy, Crohn's disease, ulcerative colitis, psoriatic arthritis, active vasculitis or gout, and siccasyndrome.
* Diagnosis of Felty Syndrome.
* Any major surgery has been performed within 8 weeks prior to the study, or will be performed during the study, from which investigators believe posing an unacceptable risk to the patient.
* Patient with cardiovascular, respiratory, liver, gastrointestinal, endocrine, hematological, neurological or psychiatric disorders or any other serious and/or unstable disease or medical history, or serious infection, and the investigators believe that these diseases or history may pose risks in the case of taking research drugs, or may interfere with the analysis of data.
* Patients who are unable to carry on normal activity or to do active work or unable to take care of themselves.
* Patients with history of malignant tumors and lymphoproliferative diseases.
* Patients with active HBV or HCV or history of HIV infection.
* Active TB diagnosed during screening or with a history of active TB that has not been appropriately treated.
* Patients who are currently pregnant or breastfeeding.
* Female patients of childbearing potential or male subjects with partners of childbearing potential not willing to use a highly effective method of contraception during the study and 28 days after last administration.
* Patient who participated in any investigational drug study within three months.

Specific laboratory abnormality including:

1. AST or ALT > 1.5 times ULN
2. Total bilirubin > 1.5 times ULN
3. Hemoglobin ≤ 85 g/L
4. White blood cells count ≤ 3.5×109/L
5. Absolute neutrophil count < 1.5×109/L
6. Lymphocyte Count < 0.75×109/L
7. Platelet count < 90×109/L
8. Creatinine > ULN

   * Any other situation, in the opinion of the investigator, characterizes the subject as not being a good candidate for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2017-03-16 (Actual); Primary Completion 2019-07-11 (Estimated); Study Completion 2019-12-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects reaching (the American College of Rheumatology response criteria 20 (ACR 20) | Week 12
  ACR 20 would be examined

SECONDARY OUTCOMES:
Change from baseline in DAS 28-CRP | Week 4/8/12
  DAS 28-CRP would be assessed
Proportion of subjects reaching ACR 20 | Week 4/8
  ACR 20 would be assessed
Proportion of subjects reaching ACR 50 and 70 | Time Frame: Week 4/8/12
  ACR 50 and 70 would be assessed
Change from baseline in ESR and CRP | Time Frame: Week 4/8/12
  ESR and CRP would assessed

CONTACTS AND LOCATIONS:
Overall Officials: Yin Su, PhD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Department of Rheumatology, Beijing, Beijing Municipality, China